CLINICAL TRIAL: NCT05626140
Title: COMPARISON OF EFFICACY OF DICLOFENAC VERSUS DICLOFENAC PLUS CODEINE AND DICLOFENAC PLUS LACOSAMIDE IN ACUTE SCIATICA
Brief Title: COMPARISON OF EFFICACY OF DIFFERENT DRUG COMBINATIONS IN ACUTE SCIATICA
Acronym: EDCLAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Collaborators: Riphah International University (Other)
Responsible Party: Principal Investigator, Dr. Mehreen Mirza, Post Graduate Trainee/ Prinicipal Investigator, Riphah International University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIMS-05-002
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Sciatica Acute; Sciatica
Keywords: Acute Sciatica, Codeine, Diclofenac, Efficacy, Lacosamide
MeSH Terms: conditions — Sciatica | interventions — Lacosamide; Tablets; Codeine; Diclofenac; dicloran

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diclofenac plus placebo (Placebo Comparator): Oral tablet diclofeanc sodium 50 mg was given with tab folic acid 5 mg as placebo ,12 hourly for 15 days
  Interventions: Drug: Diclofenac Sodium
- Diclofenac plus codeine (Active Comparator): Oral tablet diclofeanc sodium 50 mg was given with tab codeinephosphate 30 mg ,12 hourly for 15 days
  Interventions: Drug: Codeine Phosphate; Drug: Diclofenac Sodium
- Diclofenac plus lacosamide (Experimental): Oral tablet diclofeanc sodium 50 mg was given with tab lacosamide 50 mg as placebo ,12 hourly for 15 days
  Interventions: Drug: Lacosamide 50 MG Oral Tablet [Vimpat]; Drug: Diclofenac Sodium

INTERVENTIONS:
Drug: Lacosamide 50 MG Oral Tablet [Vimpat] — Oral tablet lacosamide is a 3rd generation anti convulsant drug. it is given in a dose of 50 mg 12 hourly for 15 days. It has a longer half life than the other two drugs in comparison and fewer drug interactions as it doesnot interact with the hepatic cytochrome enzymes.hence it is seen to have better pharmacokinetics and pharmacodynamics than the other drugs in study
  Other Names: Lacolap 50 mg; Vimpat 50 mg; Lalap 50 mg
  Arms: Diclofenac plus lacosamide
Drug: Codeine Phosphate — Oral Codeine Phophate is an opioid with centrally acting pain alleviating mechanisms, shorter half life and metabolized to morphine in he body which is its active metabolite
  Arms: Diclofenac plus codeine
Drug: Diclofenac Sodium — Diclofenac sodium is a Cox 2 inhibitor non steroidal anti inflammatory drug with a half life of only 1.2 hrs but a longer action of duration due to its property to get distributed to synovial fluids. metabolized to hydroxy diclofenac and excreted via urine and bile both.
  Other Names: Artifen 50 mg; Dicloran 50 mg

SUMMARY:
The goal of this clinical trial is to compare different combinations of diclofenac with diclofenac monotherapy in acute sciatica. The main questions it aims to answer are:

* Does the combination of diclofenac plus codeine better than diclofenac monotherapy for treating severe pain of sciatica
* Does the combination of diclofenac plus lacosamide better than diclofenac monotherapy for treating severe pain of sciatica

Participants will be asked to mark their pain intensity on a visual analog scale and fill oswestry disabilit index questionnaire,treatments they'll be given includes either

1. Diclofenac monotherapy
2. Diclofenac plus codeine
3. Diclofenac plus lacosamide

Researchers will compare the above three groups to see if severity of pain and disability lowered after medication

DETAILED DESCRIPTION:
Musculoskeletal conditions are the most common cause of intense long-term pain, physical disability and early deaths. They affect hundreds of millions of people of all ages irrespective of social strata globally. Lumbar radicular pain (LRP), commonly referred to as "Sciatica" is a relatively common musculoskeletal disorder.

Objective of the study is to evaluate the efficacy of different drug combinations with diclofenac for the treatment of acute sciatica. The design of the study is Single-center, clinical trial with three arms. (Single Blinding). One hundred and twenty patients were enrolled in this study between September 2021 and July 2022 at the Pharmacology department of Islamic International Medical College (IIMC) Rawalpindi in collaboration with the Neurosurgery Department, of Shaheed Zulfiqar Ali Bhutto Medical University (SZABMU) Pakistan Institute of Medical Sciences (PIMS) Islamabad. Informed verbal and written consent was taken from all patients. 40 patients were in the diclofenac (50 mg) plus placebo group, 40 in the codeine (30 mg) plus diclofenac (50 mg) group and 40 in lacosamide (50 mg) plus diclofenac (50 mg) group. Patients were followed up at day 5, 10 and 15 to assess change in pain intensity and functional disability. The use of rescue analgesia was also assessed at the final day of outcome

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute sciatica with or without lower back pain
* 18-70 years of age reporting acute pain due to sciatica

Exclusion Criteria:

* Pregnant or breastfeeding mothers.
* History of asthma or allergy to anti-inflammatory drugs.
* Mentally handicapped or terminally ill patients.
* Age less than 18 years or above 70 years
* Patients with herniated, sequestrated, or prolapsed discs waiting for surgery.
* Patient having an active ulcer (gastric or duodenal) or bleeding from the stomach or bowel.
* Patients already taking an anti-depressant medication, a medication for neuropathic pain, an anticonvulsant, or a sedative and unable to cease the medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Patients were asked to mark a line and record their pain scores at baseline and day 5, day 10 and day 15
  Severity of leg pain or lower back pain associated with acute sciatica to be assessed using the visual analog scale VAS to determine if the mean pain scores decreased during the course of the medication. VAS is a commonly used pain score in interventinal studies and evaluating pain intensity related with musculoskeletal disorders or post opertive types of pain. For this , the patient is asked to mark a line anywhere on a 10 cm line with 0 taken on the left edge. The mark drawn on the line corresponds to the intensity pf pain experienced by the patient at the time of the pain assessment

SECONDARY OUTCOMES:
Functional Disbability | ODI was measured at baseline and days 5,10, and 15 and patients were asked to fill the questionnaire on the respective days
  The ODI is an index derived from the Oswestry Low Back Pain Questionnaire. The self-administered questionnaire consists of ten topics related to intensity of pain, lifting, ability of self-care, potential to walk, capacity to sit, sexual function, strength to stand, social life, quality of sleep, and capability to travel. Each category (topic) is then followed by 6 statements relating different potential scenarios in the patient's life concerning to the topic. Patients are inquired to specify the statement that most strictly is similar to their situation. Statements are linked with scores from 0 to 5, where 0 represents the lowest disability and 5 equivalent to extreme disability. The sum of the ten scores is stated as a percentage of the maximum score (50) ranging from 0% = no disability to 100% = maximum disability

OTHER OUTCOMES:
Use of Rescue Analgesia | The use of rescue medication was determined on the final day of outcome i.e. Day 15
  This parameter was evaluated if the patient used rescue medication (YES or NO) in case the pain did not improve or settle with the medicines already given to the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Mehreen Mirza, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No